CLINICAL TRIAL: NCT03949751
Title: Can Propionibacterium Acnes Load in Primary Shoulder Surgery be Reduced With Preoperative Application of a Benzoylperoxid/Miconazolnitrat crème Additional to Standard Antibiotic Prophylaxis
Brief Title: Acne crème to Reduce Propionibacterium Acnes Load in Primary Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W728
Record Dates: First submitted 2019-02-15; First posted 2019-05-14 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Shoulder Infections
Keywords: gram positive bacteria; Benzoylperoxid and Miconazolnitrat

STUDY DESIGN:
Intervention Model Description: 30 patients will get Acne Crème Plus (Benzoylperoxid and Miconazolnitrat) to apply until operation (on average 7 days) after receiving written consent. The application should be done daily in the evening on the planned operative side covering the skin from the nipple-areola complex laterally to the medial margin of the scapula and from a horizontal line through the nipple-areola complex cranially over the shoulder and dorsally to the spina scapulae. 30 patients will be included in the control group. Those patients will not get the local therapy in the preoperative consultation but they will need to give written consent for taking swabs for culture samples pre- and intraoperative.
Who Masked: Investigator
Masking Description: The institution has a standardized procedure for recruiting participants as participant studies are common. They will be preselected, based on the in- and exclusion criteria as mentioned above. If the match the inclusion criteria and do not meet the exclusion criteria, they will be informed, during the preoperative consultation by one of the study investigators, about the study, its nature, purpose, procedures involved, expected duration, participating investigators, potential risks and benefits and any potential discomfort the study could entail. The first 30 patients that can be selected through this procedure for the participation in the study will not get any therapy and therefore they will form the control group. The next 30 patients will get the therapy and so form the treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The participants of the control group will not get the local therapy in the investigator's preoperative consultation but they will need to give written consent for taking swabs for culture samples pre- and intraoperative.
- Therapy group (Experimental): 30 patients will get Acne Crème Plus (Benzoylperoxid and Miconazolnitrat) to apply until operation (on average 7 days) after receiving written consent. The application should be done daily in the evening on the planned operative side covering the skin from the nipple-areola complex laterally to the medial margin of the scapula and from a horizontal line through the nipple-areola complex cranially over the shoulder and dorsally to the spina scapulae.
  Interventions: Drug: Acne Crème Plus

INTERVENTIONS:
Drug: Acne Crème Plus — The study specific intervention product is a combination of Benzoylperoxid and Miconazolnitrat (Widmer Acne Crème Plus, 47033 Swissmedic) to apply daily in the evening on the skin from the nipple-areola complex laterally to the medial margin of the scapula and from a horizontal line through the nipple-areola complex cranially over the shoulder and dorsally to the spina scapulae. The application should be done regularly for 7 days before shoulder surgery. The study specific intervention product is authorized by Swissmedic for use in the treatment of acne and is used standardly in clinical practice.
  Other Names: Widmer Acne Crème Plus, 47033 (Swissmedic)
  Arms: Therapy group

SUMMARY:
60 patients undergoing first time open shoulder surgery (Latarjet, prosthesis) will be prospectively included in this study. The investigators will do a randomized controlled trial, choosing with a single-blinded protocol 30 patients for local therapy and other 30 patients as the control group without any treatment preoperative. In the preoperative consultation 30 patients will get Acne Crème Plus (Benzoylperoxid and Miconazolnitrat) to apply until operation (on average 7 days) after receiving written consent. The application should be done daily in the evening on the planned operative side covering the skin from the nipple-areola complex laterally to the medial margin of the scapula and from a horizontal line through the nipple-areola complex cranially over the shoulder and dorsally to the spina scapulae. 30 patients will be included in the control group. Those patients will not get the local therapy in the preoperative consultation but they will need to give written consent for taking swabs for culture samples pre- and intraoperative. In the operation room there will be done from each of the 60 patients a superficial skin swab before doing disinfection, a swab of the subcutaneous layer and a swab of the deep layer (joint capsule). All the three swabs from each of the 60 patients will be sent to Unilabs, Labor für Medizinische Analytik AG, Dübendorf, Switzerland to streak on agar plates to cultivate under anaerobic conditions for 14 days. Propionibacterium acnes will be identified by use of matrix-assisted laser desorption/ionization time-of-flight mass spectrometry.

DETAILED DESCRIPTION:
According to recent studies, Propionibacterium acnes is found in 30% of patients with no preliminary shoulder operation and without obvious signs of infection. This bacterium is supposed to be the main pathogen causing shoulder infections. As it resides in the subcutaneous layer, many antiseptic and antibiotic agents that affect other layers fail to prevent infections. When administering antibiotics to reduce infections due to Propionibacterium acnes, cross-resistances to various antibiotics are created. Therefore, the investigators aim to investigate the efficacy of a local combination therapy without antibiotics (Benzoylperoxid and Miconazolnitrat) to reduce the presence of Propionibacterium acnes in patients first time undergoing open shoulder surgery. The investigators will also demonstrate the rate of positive cultures for Propionibacterium acnes in different layers regarding gender and age of patients. To best knowledge, no randomized controlled trials investigating the efficacy of Benzoylperoxid and Miconazolnitrat for reduction of Propionibacterium acnes in patients undergoing first time open shoulder surgery exist in the literature. However, in 1989 a clinical trial could demonstrate a 66% reduction of inflammatory acne lesions by applying a lotion containing Benzoylperoxid and Miconazol.

The investigators suppose that the patients with the local therapy (therapy group) show fewer positive samples than the patients of the control group as the combination of Benzoylperoxid and Miconazolnitrat (Widmer Acne Crème Plus, approval number 47033, Swissmedic) is used in the therapy of acne where Propionibacterium acnes is the major pathogen. By decreasing the presence of Propionibacterium acnes, infections and revision surgeries could be reduced as well. The investigators expect a higher rate of positive cultures from the subcutaneous layer compared to the superficial and to the deep layer. The investigators await more positive cultures in men than in women as men show a higher density of the glands in the subcutaneous layer where Propionibacterium acnes is linked to. For the same reason, the investigators suppose also a higher number of positive culture samples in younger patients (≤40 years) than in older patients (>40 years).

60 patients undergoing first time open shoulder surgery (Latarjet, prosthesis) will be prospectively included in this study. The investigators will do a randomized controlled trial, choosing with a single-blinded protocol 30 patients for local therapy and other 30 patients as the control group without any treatment preoperative. In the preoperative consultation 30 patients will get Acne Crème Plus (Benzoylperoxid and Miconazolnitrat) to apply until operation (on average 7 days) after receiving written consent. The application should be done daily in the evening on the planned operative side covering the skin from the nipple-areola complex laterally to the medial margin of the scapula and from a horizontal line through the nipple-areola complex cranially over the shoulder and dorsally to the spina scapulae. 30 patients will be included in the control group. Those patients will not get the local therapy in the preoperative consultation but they will need to give written consent for taking swabs for culture samples pre- and intraoperative. In the operation room there will be done from each of the 60 patients a superficial skin swab before doing disinfection, a swab of the subcutaneous layer and a swab of the deep layer (joint capsule). All the three swabs from each of the 60 patients will be sent to Unilabs, Labor für Medizinische Analytik AG, Dübendorf, Switzerland to streak on agar plates to cultivate under anaerobic conditions for 14 days. Propionibacterium acnes will be identified by use of matrix-assisted laser desorption/ionization time-of-flight mass spectrometry. The number of positive culture samples from the therapy group will be compared with the number of positive culture samples from the control group.

Determination of Sample Size was done by performing a power analysis using www.clincalc.com, a sample size calculator placed at disposal by Sean P. Kane (clinical pharmacist, assistant professor at Rosalind Franklin University of Medicine and Science, North Chicago and advocate of evidence-based medicine). The study groups are two independent groups as they receive different treatments. The primary endpoint is dichotomous. The anticipated incidence of the therapy group is defined as 30%, the incidence of the control group is supposed to be 3-5% and the enrolment ratio is 1. The probability of a type-I-error is 0.05. With obtaining a power of 80%, between 56 and 70 participants are needed for the study according to the sample size calculator.

Recent studies could show that 30% of the patients without any obvious signs for infection and no preliminary operation have positive culture samples for Propionibacterium acnes, the investigators expect this result as well. The investigators suppose that the patients with the local therapy (therapy group) show fewer positive samples than the patients of the control group as the combination of Benzoylperoxid and Miconazolnitrat is used in the therapy of acne where Propionibacterium acnes is the major pathogen. As it is known that Propionibacterium acnes resides in the subcutaneous layer, the investigators expect a higher rate of positive cultures from the subcutaneous layer compared to the superficial and to the deep layer. The investigators expect more positive cultures in men than in women as men show a higher density of the glands in the subcutaneous layer where Propionibacterium acnes is linked to. The investigators suppose also a higher number of positive culture samples in younger patients (≤40 years) than in older patients (>40 years).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing first time open shoulder surgery (Latarjet, prosthesis)
* Male and female patients
* Age > 18 years
* Competent German language skills
* Written informed consent as documented by signature (Appendix Informed Consent Form)

Exclusion Criteria:

* Previous enrollment into the current study,
* known or suspected non-compliance, drug or alcohol abuse,
* participation in another study with investigational drug within the 30 days preceding and during the present study,
* pregnancy or breast feeding (see chapter 3.7),
* preliminary shoulder surgeries,
* patients planned for an arthroscopic shoulder surgery,
* hypersensitivity to Benzoylperoxid or Miconazol,
* use of other acne preparations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-05-23 (Actual)

PRIMARY OUTCOMES:
Positive Propionibacterium acnes sample therapy group before therapy | 1 day
  Number of positive culture samples for Propionibacterium acnes in patients undergoing first time open shoulder surgery in the therapy group at the time point before application of therapy.
Positive Propionibacterium acnes sample control group before surgery | 1 day
  Number of positive culture samples for Propionibacterium acnes in patients undergoing first time open shoulder surgery in the control group at the time point before application of therapy in the therapy Group.
Change of positive Propionibacterium acnes sample therapy group after therapy | Around 7 days
  Number of positive culture samples for Propionibacterium acnes in patients undergoing first time open shoulder surgery in the therapy group after application of therapy.
Change of positive Propionibacterium acnes sample control group intraoperative | Around 7 days
  Number of positive culture samples for Propionibacterium acnes in patients undergoing first time open shoulder surgery in the control group after application of therapy in the therapy group.

SECONDARY OUTCOMES:
Change of positive Propionibacterium acnes in different layers | Around 7 days
  Rate of positive cultures for Propionibacterium acnes in different layers (superficial, subcutaneous, deep layer)
Change of positive Propionibacterium acnes gender-related | Around 7 days
  Rate of positive cultures for Propionibacterium acnes in male versus female
Change of positive Propionibacterium acnes age-related | Around 7 days
  Rate of positive cultures for Propionibacterium acnes in younger versus older patients

CONTACTS AND LOCATIONS:
Overall Officials: Samy Bouaicha, PD Dr.med., Principal Investigator — Balgrist University Hospital
Locations (1):
- University Hospital Balgrist, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD.

REFERENCES:
- [Background] Padegimas EM, Lawrence C, Narzikul AC, Zmistowski BM, Abboud JA, Williams GR, Namdari S. Future surgery after revision shoulder arthroplasty: the impact of unexpected positive cultures. J Shoulder Elbow Surg. 2017 Jun;26(6):975-981. doi: 10.1016/j.jse.2016.10.023. Epub 2017 Jan 10. PMID 28087166
- [Background] Achermann Y, Sahin F, Schwyzer HK, Kolling C, Wust J, Vogt M. Characteristics and outcome of 16 periprosthetic shoulder joint infections. Infection. 2013 Jun;41(3):613-20. doi: 10.1007/s15010-012-0360-4. Epub 2012 Nov 3. PMID 23124880
- [Background] Levy O, Iyer S, Atoun E, Peter N, Hous N, Cash D, Musa F, Narvani AA. Propionibacterium acnes: an underestimated etiology in the pathogenesis of osteoarthritis? J Shoulder Elbow Surg. 2013 Apr;22(4):505-11. doi: 10.1016/j.jse.2012.07.007. Epub 2012 Sep 13. PMID 22981447
- [Background] Dodson CC, Craig EV, Cordasco FA, Dines DM, Dines JS, Dicarlo E, Brause BD, Warren RF. Propionibacterium acnes infection after shoulder arthroplasty: a diagnostic challenge. J Shoulder Elbow Surg. 2010 Mar;19(2):303-7. doi: 10.1016/j.jse.2009.07.065. Epub 2009 Nov 1. PMID 19884021
- [Background] Phadnis J, Gordon D, Krishnan J, Bain GI. Frequent isolation of Propionibacterium acnes from the shoulder dermis despite skin preparation and prophylactic antibiotics. J Shoulder Elbow Surg. 2016 Feb;25(2):304-10. doi: 10.1016/j.jse.2015.08.002. Epub 2015 Oct 9. PMID 26456428